CLINICAL TRIAL: NCT02448927
Title: The preDIlatation in tRanscathEter aortiC Valve implanTation Trial
Acronym: DIRECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Konstantinos Toutouzas, Associate Professor of Cardiology, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIRECT Trial
Record Dates: First submitted 2015-01-14; First posted 2015-05-20 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Aortic Valve Stenosis
Keywords: transcatheter aortic valve implantation; Balloon aortic valvuloplasty; Aortic stenosis; TAVI; TAVR (transcatheter aortic valve replacement); CoreValve; BAV; Evolut R
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAVI patients without balloon aortic valvuloplasty (Other): Patients that will not undergo balloon aortic valvuloplasty (BAV) before transcatheter aortic valve intervention (TAVI) with the Medtronic Evolut R (or CoreValve).
  Interventions: Device: Transcatheter Aortic Valve Implantation
- TAVI patients with balloon aortic valvuloplasty (Active Comparator): Patients that will undergo balloon aortic valvuloplasty (BAV) before transcatheter aortic valve intervention (TAVI) with the Medtronic Evolut R (or CoreValve).
  Interventions: Device: balloon aortic valvuloplasty; Device: Transcatheter Aortic Valve Implantation

INTERVENTIONS:
Device: balloon aortic valvuloplasty
  Other Names: BAV
  Arms: TAVI patients with balloon aortic valvuloplasty
Device: Transcatheter Aortic Valve Implantation
  Other Names: TAVI

SUMMARY:
This is a randomized trial that will evaluate the role of balloon aortic valvuloplasty (BAV) on the outcome of patients undergoing transcatheter aortic valve implantation (TAVI) procedure. Patients will undergo a physical exam, coronary angiography and computed tomography angiography before TAVI. The randomization for direct or non-direct TAVI ( with BAV or without BAV) will take place 24 hours prior to the procedure by the core lab at Hippokration Hospital in Athens. The same lab will analyze in blind fashion the results of all the imaging modalities for each patient. The patients will be followed during the hospital stay and at 30 days and 1 year thereafter by echocardiography. The procedure of predilatation will be at the operator's discretion.

DETAILED DESCRIPTION:
Background: Balloon aortic valvuloplasty (BAV) is a vital part of the transcatheter aortic valve implantation (TAVI) procedure. There is a lack of long-term evidence in patients undergoing direct TAVI without predilatation.

Trial: This is a prospective multi-center randomized trial.

Participating medical centers:

1. 1st Department of Cardiology, Hippokration Hospital/Athens Medical School, Athens, Greece
2. Heart Institute, Hadassah Hebrew University Medical Center, POB 12000, Jerusalem 91120, Israel.
3. Department of Cardiology, Division of Internal Medicine, University Medical Centre Ljubljana, Zaloška 7, SI-1525 Ljubljana, Slovenia.
4. Department of Cardiology, Onassis Cardiac Surgery Center, Athens, Greece
5. Second Department of Cardiology, University Hospital of Ioannina, Ioannina, Greece

Description: Patients will undergo a physical exam, coronary angiography and computed tomography angiography before TAVI. The randomization for direct or non-direct TAVI will take place 24 hours prior to the procedure by the core lab at Hippokration Hospital in Athens. The same lab will analyze in blind fashion the results of all the imaging modalities for each patient. The patients will be followed during the hospital stay and at 30 days and 1 year thereafter by echocardiography. The procedure of predilatation will be at the operator's discretion. Access sites for TAVI are: transfemoral, subclavian and transaortic.

ELIGIBILITY:
Inclusion Criteria:

1. Diameter of >5mm for Evolut R and >6mm for CoreValve of the vessel.
2. Aortic valve diameter of ≥20mm and ≤29mm as measured by echo.
3. Ascending aorta diameter ≤ 43mm at the sinotubular junction.
4. Severe aortic stenosis, defined as aortic valve area of < 1.0 cm2 (or aortic valve area index of < 0.6 cm2/m2) by the continuity equation, AND mean gradient > 40 mmHg or maximal aortic valve velocity > 4.0 m/sec by resting echocardiogram.
5. STS score of ≥ 8 OR LogEuroSCORE> 20%, OR

   * 80 years old OR
   * 65 years old with 1 or 2 (but not more than two) from the following criteria:

     * Liver cirrhosis (Class A or B).
     * Pulmonary insufficiency: VMS<1 liter.
     * Previous heart surgery (CABG, vascular surgery).
     * Porcelain aorta.
     * Pulmonary artery systolic pressure >60 mmHg and high risk for heart surgery.
     * Relapsing pulmonary embolism.
     * Right ventricular insufficiency.
     * Thoracic wall injuries that contraindicate an open heart surgery.
     * History of radiation therapy of the mediastinum.
     * Connective tissue disease that contraindicates an open heart surgery.
     * Frailty/cachexia.
6. Patients will be informed on the nature of the study and provide written consent.

Exclusion Criteria:

1. A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated: aspirin or heparin and bivalirudin, ticlopidine and clopidogrel, nitinol (titanium or nickel), contrast media
2. Ongoing sepsis, including active endocarditis.
3. Any percutaneous coronary or peripheral interventional procedure with a bare metal or drug eluting stent performed within 30 days prior to Heart Team assessment.
4. Echocardiographic evidence of LV or LA thrombus.
5. Mitral or tricuspid valve insufficiency (> grade II).
6. Previous aortic valve replacement (mechanical or bioprosthetic).
7. Recent (within 6 months of Heart Team assessment) cerebrovascular accident (CVA) or transient ischemic attack (TIA).
8. Patients with:

   Femoral, iliac or aortic vascular disease (stenosis etc) that precludes the insertion of a transcatheter sheath.

   OR Symptomatic carotid or vertebral artery disease (> 70% stenosis).
9. The patient has a bleeding diathesis, coagulopathy or denies blood transfusion.
10. Estimated life expectancy of less than 12 months due to associated non-cardiac co-morbid conditions.
11. Creatinine clearance < 20 ml/min.
12. Active gastritis or ulcer.
13. Pregnancy.
14. Severe left ventricular dysfunction with left ventricular ejection fraction (LVEF) < 20%.
15. Unicuspid or bicuspid aortic valve.
16. Mixed aortic valve disease (aortic stenosis and aortic regurgitation> 2+).
17. Liver failure (Child-Pugh class C).
18. Severe dementia (resulting in either inability to provide informed consent for the study/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits).
19. Extreme aortic valve calcification and calcific asymmetry (if semiquantitively measured: grade 4, Agatston score: grade 4 AgS>5000 AU).
20. Aortic valve area of < 0.4 cm2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2015-05; Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Device success | 30 days
  Device success, as designated by the VARC-2 criteria.

SECONDARY OUTCOMES:
Death | 30 days
  Death during the hospitalization of the patient, as designated by the VARC-2 criteria.
Cerebrovascular accident | 30 days and 1 year
  Cerebrovascular accident during and after the hospitalization of the patient, as designated by the VARC-2 criteria.
New pacemaker implantation | 30 days
  New pacemaker implantation during the hospitalization of the patient, as designated by the VARC-2 criteria.
Vascular complications | 30 days
  Vascular complications during the hospitalization of the patient, as designated by the VARC-2 criteria.
Mortality | after 30 days and at 1 year
  Death after discharge of the patient, as designated by the VARC-2 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Tousoulis, Professor, Study Chair — University of Athens
Locations (4):
- Greece (3):
  - First Department of Cardiology, University of Athens, Athens, Attica
  - Department of Cardiology, Onassis Cardiac Surgery Center, Athens
  - Second Department of Cardiology, University Hospital of Ioannina, Ioannina
- Heart Institute Hadassah Hebrew University Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Toutouzas K, Benetos G, Voudris V, Drakopoulou M, Stathogiannis K, Latsios G, Synetos A, Antonopoulos A, Kosmas E, Iakovou I, Katsimagklis G, Mastrokostopoulos A, Moraitis S, Zeniou V, Danenberg H, Vavuranakis M, Tousoulis D. Pre-Dilatation Versus No Pre-Dilatation for Implantation of a Self-Expanding Valve in All Comers Undergoing TAVR: The DIRECT Trial. JACC Cardiovasc Interv. 2019 Apr 22;12(8):767-777. doi: 10.1016/j.jcin.2019.02.005. Epub 2019 Mar 27. PMID 30928442